CLINICAL TRIAL: NCT06434935
Title: Initial Evaluation of Vascudyne Coronary Artery Bypass Conduit
Acronym: VCAB-1
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vascudyne, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-003
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: CABG; Coronary bypass
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- True CABA (Experimental): Patients will be implanted with a single TRUE CAB bypass (single proximal and distal anastomoses) to the second or third CA bypass target
  Interventions: Combination Product: CABA

INTERVENTIONS:
Combination Product: CABA — Coronary Bypass

SUMMARY:
The Vascudyne Coronary Artery Bypass Study (VCAB-1) is an initial safety and feasibility study of the Vascudyne, Inc. Coronary Artery Bypass Conduit (CAB A) for bypass of stenosed native coronary arteries in patients undergoing coronary artery bypass surgery.

DETAILED DESCRIPTION:
Prospective, non-randomized, initial evaluation clinical study to assess the feasibility of TRUE CAB for secondary coronary targets in patients needing multiple coronary artery bypass.

Patients will be implanted with a single TRUE CAB bypass (single proximal and distal anastomoses) to the second or third coronary arteries (CA) bypass target.

The primary target CA shall be bypassed using an arterial graft. The left anterior descending (LAD) CA bypass, if needed, shall be bypassed using the left internal mammary artery (LIMA). A saphenous vein shall be used for any additional targets as needed.

Estimated enrollment for first three patients (2 weeks), followed by enrollment over 4 months. Follow up through 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients needing isolated coronary artery bypass grafting to multiple coronary arteries (CA) in which the first target CA shall be an arterial bypass to the left anterior descending artery (LAD) and the second and potentially third target CA must be at least 2 mm in diameter, have at least 70% stenosis proximal to the bypass, have at least Thrombolysis in Myocardial Infarction (TIMI) II flow, and shall be among the following options: right coronary artery (RCA), right posterior descending artery (PDA), Ramus Intermedius, obtuse marginal arteries (OM), or diagonal branches of the left anterior descending artery.
2. Male or female patients between the ages of 45 and 75 years inclusive.
3. Elective patient, selected and accepted by the local Heart Team and confirmed by the Sponsor's Screening Committee for an on-pump full sternotomy CABG surgery.
4. Life expectancy of at least 4 years.
5. Female subjects must be of non-childbearing potential, which is defined as post-menopausal (at least 1 year without menses prior to Screening) or documented surgically sterile or post hysterectomy (at least 1 month prior to Screening).
6. Patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.
7. Patient has been informed and agrees to pre- and post-procedure follow-up, including follow-up cardiac ultrasound and coronary angiogram or computerized tomography (CT) scan.
8. Patient is willing to be compliant with prescribed anticoagulant therapy (critical to preventing thrombus in the investigational device).

Exclusion Criteria:

1. Patients with left ventricular ejection fraction < 35%.
2. Patients with diffusely diseased coronary arteries suggestive of either poor target quality, or poor vessel runoff.
3. Patients requiring emergency surgery.
4. Patients with cardiogenic shock.
5. Patients with any prior open cardiac surgery such as coronary artery bypass graft (CABG).
6. Any planned concomitant cardiac surgery, including but not limited to: valve surgery, repair of intracardiac shunt, surgical arrhythmia ablation.
7. History of cardiac resynchronization therapy (CRT) or implantable cardioverter defibrillator (ICD) implantation.
8. Myocardial infarction (MI) within 21 days or cerebral vascular accident (CVA) within 90 days of the CABG procedure.
9. Patients with Type 1 Diabetes and Patients with Type II Diabetes having glycate hemoglobin test (A1C)>8.
10. Chronic kidney disease with Glomerular Filtration Rate (GFR) < 45 militers per minute (mL/min), or active dialysis patients
11. Moderate to severe chronic obstructive pulmonary disease (COPD) with a forced expiratory volume (FEV) <1.5 lit/sec or 45% predicted forced expiratory volume in one second (FEV1).
12. Patient with known interstitial lung disease, diagnosed by imaging or pulmonary function tests, including diffusing capacity of the lungs for carbon monoxide (DLCO).
13. Endocarditis, pericarditis, or any other active systemic infection that would interfere with patient safety.
14. Patient on preoperative anticoagulant (i.e. Warfarin) or any known intrinsic coagulation disorder.
15. Abnormal blood values (e.g. leukopenia, anemia, thrombocytopenia, or thrombocytosis with Platelet Count >400,000 per militer (mL) that could influence graft hemostasis or patient recovery.
16. Known allergies to study device components: Nitinol, Nickel, Titanium, or agents/medication such as contrast agents, antiplatelet therapy, beta-blocker, or statins required for study assessment or optimal post-CABG medical treatment (hospital standard of care).
17. Any medical intervention or condition within the 12 months following TRUE CAB implantation that requires temporary or permanent discontinuation of anticoagulant therapy.
18. History of heparin-induced thrombocytopenia.
19. Contraindication to or known serious allergy to anticoagulant, aspirin, or planned antiplatelet and factor Xa inhibitor therapy.
20. Immunodeficiency including AIDS / HIV, active autoimmune disease, or on immunosuppressant therapy.
21. Treatment with any investigational drug or device within 60 days prior to study entry or ongoing participation in another clinical study of an investigational product.
22. Subject has medical, social, or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance.
23. Has any other condition, in the opinion of the principal investigator, which would put the patient at increased risk from participating in the study or otherwise prevent participation.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Patency | 6 months
  Intervention-free angiographic patency [failure defined as >50% stenosis or occlusion].
Major Adverse Cardiac and Cerebrovascular events (MACCE) | 30 days
  Freedom from MACCE; includes adverse events; death, non-fatal myocardial infraction, non-fatal stroke, unplanned revascularization, and hospitalization due to heart failure

SECONDARY OUTCOMES:
Patency | 30 days, 12 months, 18 months and 24 months
  Intervention-free angiographic patency [failure defined as >50% stenosis or occlusion].
Fitzgibbon classification | 30 days, 6 months and 12 months
  Fitzgibbon classification is a grading system for coronary artery bypass grafts (CABGs) that use saphenous vein grafts (SVGs) and arterial grafts to treat severe coronary artery disease. The scale assesses the following characteristics:
  Fitzgibbon I patency (perfect patency) with no lumen irregularities. Fitzgibbon II patency with lumen irregularities that involve less than 50% of SVG length.
  Fitzgibbon III patency with lumen irregularities that involve more than 50% of SVG length
MACCE | 6, 12, 18 and 24 months
  Freedom from MACCE includes adverse events; death, non-fatal myocardial infraction, non-fatal stroke, unplanned revascularization, and hospitalization due to heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ebner, MD, Principal Investigator — Italian Hospital Asuncion Paraguay
Locations (1):
- Sanatario Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No